CLINICAL TRIAL: NCT02057692
Title: The Evaluation of the Intestinal Bile Acid Transport (IBAT) Inhibitor LUM001 in the Reduction of Pruritus in Alagille Syndrome, a Cholestatic Liver Disease
Brief Title: Evaluation of LUM001 in the Reduction of Pruritus in Alagille Syndrome
Acronym: ITCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Collaborators: Childhood Liver Disease Research and Education Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LUM001-301; NCT02055768 (obsolete NCT alias)
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Alagille Syndrome
MeSH Terms: conditions — Alagille Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LUM001 (Experimental): LUM001 for oral administration
  Interventions: Drug: LUM001
- Placebo (Placebo Comparator): Placebo administered orally once each day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LUM001 — LUM001 administered orally
  Arms: LUM001
Drug: Placebo — Placebo administered orally
  Arms: Placebo

SUMMARY:
The study is a randomized, double-blind, placebo-controlled study in children with Alagille Syndrome (ALGS). The study will investigate the effects of LUM001, compared to placebo, on pruritus, serum bile acids, liver enzymes, and other biochemical markers in patients with ALGS.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Alagille Syndrome
2. Evidence of cholestasis
3. Moderate to severe pruritus
4. Ability to understand and willingness to sign informed consent/assent prior to initiation of any study procedures

Exclusion Criteria:

1. Surgical disruption of the enterohepatic circulation
2. Liver transplant
3. History or presence of other concomitant liver disease
4. Females who are pregnant or lactating
5. Known HIV infection

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mirum
Locations (13):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 13 study centers in the United States and Canada, between 24 November 2014 (first participant first visit) and 16 November 2016 (last participant last visit).
Pre-assignment Details: Overall, 37 participants were enrolled to dose escalation phase started with 14 microgram per kilogram per day (mcg/kg/day) per week on Week 1 up to 280 mcg/kg/day for a maximum up to 5 weeks, until they reached the planned stable dose of 70, 140 and 280 mcg/kg/day and continued up to Week 13.
Groups:
- Maralixibat 70 mcg/kg/Day: Participants received low dose maralixibat 70 mcg/kg/day oral solution for 10 weeks during the stable dosing period, which was administered after a dose escalation period, in which participants received 14, 35 and 70 mcg/kg/day dose per each week respectively up to 3 weeks.
- Maralixibat 140 mcg/kg/Day: Participants received mid dose maralixibat 140 mcg/kg/day oral solution for 9 weeks during the stable dosing period, which was administered after a dose escalation period, in which participants received 14, 35, 70 and 140 mcg/kg/day dose per each week respectively up to 4 weeks.
- Maralixibat 280 mcg/kg/Day: Participants received high dose maralixibat 280 mcg/kg/day oral solution for 8 weeks during the stable dosing period, which was administered after a dose escalation period, in which participants received 14, 35, 70, 140 and 280 mcg/kg/day dose per each week respectively up to 5 weeks.
- Placebo: Participants received placebo matched to maralixibat oral solution for 13 weeks (dose escalation and stable dosing period).
Period: Overall Study
Arm/Group | Maralixibat 70 mcg/kg/Day | Maralixibat 140 mcg/kg/Day | Maralixibat 280 mcg/kg/Day | Placebo
Started | 8 | 11 | 6 | 12
Completed | 7 | 11 | 6 | 11
Not Completed | 1 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population included all participants who were randomly assigned to study treatment and received at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Maralixibat 70 mcg/kg/Day | Maralixibat 140 mcg/kg/Day | Maralixibat 280 mcg/kg/Day | Placebo | Total
Number analyzed (Participants) | 8 | 11 | 6 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.4 (4.75) | 8.6 (4.32) | 5.5 (4.76) | 5.5 (4.19) | 6.8 (4.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 6 | 16
  Male | 6 | 7 | 2 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint (Week 13/Early Termination) in Pruritus
Description: Pruritus was assessed using Itch report outcome measure (ItchRO[Obs]), administered as an electronic diary (eDiary) which was completed by the participants twice daily (morning and evening). ItchRO(Obs) score ranged from 0 to 4, with the higher score indicating increasing itch severity. The highest score between the morning and evening ItchRO(Obs) reports represented the daily score: a measure of the worst itching over the previous 24-hour period.
Time Frame: Baseline, Week 13/Early Termination
Population: Modified Intent-to-Treat Population (mITT) population included all participants randomly assigned to study treatment, receiving at least 1 dose of treatment, and having at least 1 post baseline observer itch reported outcome (ItchRO[Obs]) average daily score.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Maralixibat 70 mcg/kg/Day | Maralixibat 140 mcg/kg/Day | Maralixibat 280 mcg/kg/Day | Placebo
Number analyzed (Participants) | 8 | 11 | 6 | 12
Score on a scale | -1.470 (0.3034) | -1.486 (0.2597) | -0.620 (0.3575) | -0.580 (0.2453)
Statistical Analysis 1: Comparison: Maralixibat 70 mcg/kg/Day vs Placebo; The primary analysis of change from baseline to endpoint (Week 13/ET) average daily ItchRO(Obs) was evaluated by analysis of covariance (ANCOVA) using a PROC MIXED procedure. Least-squares (LS) mean change from baseline to Endpoint (Week 13/ET), along with associated 95% confidence interval (CI) for the LS mean, and pair-wise treatment P-values were calculated for each treatment group; Test type: Superiority; p = 0.0321, ANCOVA; LS mean difference = -0.889, 95% CI 2-sided [-1.698 to 0.081], Standard Error of Mean 0.3969
Statistical Analysis 2: Comparison: Maralixibat 140 mcg/kg/Day vs Placebo; The primary analysis of change from baseline to endpoint (Week 13/ET) average daily ItchRO(Obs) was evaluated by ANCOVA using a PROC MIXED procedure. LS mean change from baseline to Endpoint (Week 13/ET), along with associated 95% CI for the LS mean, and pair-wise treatment P-values were calculated for each treatment group; Test type: Superiority; p = 0.0145, ANCOVA; LS mean difference = -0.906, 95% CI 2-sided [-1.620 to -0.192], Standard Error of Mean 0.3503
Statistical Analysis 3: Comparison: Maralixibat 280 mcg/kg/Day vs Placebo; The primary analysis of change from baseline to endpoint (Week 13/ET) average daily ItchRO(Obs) was evaluated by ANCOVA using a PROC MIXED procedure. LS mean change from baseline to Endpoint (Week 13/ET), along with associated 95% confidence interval (CI) for the LS mean, and pair-wise treatment P-values were calculated for each treatment group; Test type: Superiority; p = 0.9298, ANCOVA; LS mean difference = -0.039, 95% CI 2-sided [-0.942 to 0.863], Standard Error of Mean 0.4431

2. Secondary Outcome: Change From Baseline to Endpoint (Week 13/Early Termination) in Fasting Serum Bile Acid (sBA) Level
Description: Fasting sBA level was measured by using a liquid chromatography mass spectrometry method.
Time Frame: Baseline, Week 13/Early Termination
Population: mITT population included all participants randomly assigned to study treatment, receiving at least 1 dose of treatment, and having at least 1 post baseline observer itch reported outcome (ItchRO[Obs]) average daily score.
Measure: Least Squares Mean (Standard Error); unit: Micro moles per liter (mcmol/L)
Arm/Group | Maralixibat 70 mcg/kg/Day | Maralixibat 140 mcg/kg/Day | Maralixibat 280 mcg/kg/Day | Placebo
Number analyzed (Participants) | 8 | 11 | 6 | 12
Micro moles per liter (mcmol/L) | -117.401 (46.2353) | -40.358 (34.8650) | -27.437 (46.2823) | -10.442 (32.6776)

3. Secondary Outcome: Change From Baseline to Endpoint (Week 13/Early Termination) in Liver Enzyme Levels
Description: Liver enzyme levels of alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase and gamma glutamyl transferase were reported here.
Time Frame: Baseline, Week 13/Early Termination
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Unit per liter (U/L)
Arm/Group | Maralixibat 70 mcg/kg/Day | Maralixibat 140 mcg/kg/Day | Maralixibat 280 mcg/kg/Day | Placebo
Number analyzed (Participants) | 8 | 11 | 6 | 12
Unit per liter (U/L)
  Alanine Aminotransferase | 14.616 (17.9442) | 13.236 (14.9424) | 29.539 (19.6083) | -11.928 (13.9736)
  Alkaline Phosphatase | 46.276 (38.9056) | -9.570 (30.8065) | -3.280 (42.1582) | 32.502 (29.9885)
  Aspartate Aminotransferase | 20.241 (16.8467) | 11.851 (13.9367) | 16.539 (18.3472) | -3.691 (13.0114)
  Gamma Glutamyl Transferase | -48.124 (46.2867) | 48.053 (36.1507) | -10.937 (48.8614) | -37.757 (34.7766)

4. Secondary Outcome: Change From Baseline to Endpoint (Week 13/Early Termination) in Total and Direct Bilirubin Concentrations
Description: Liver enzyme levels of total bilirubin and direct bilirubin were reported here.
Time Frame: Baseline, Week 13/Early Termination
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Maralixibat 70 mcg/kg/Day | Maralixibat 140 mcg/kg/Day | Maralixibat 280 mcg/kg/Day | Placebo
Number analyzed (Participants) | 8 | 11 | 6 | 12
Milligrams per deciliter (mg/dL)
  Total Bilirubin | -0.291 (0.3777) | -0.353 (0.3014) | -0.804 (0.4021) | 0.104 (0.2847)
  Direct Bilirubin | -0.333 (0.2086) | -0.305 (0.1672) | -0.508 (0.2243) | 0.011 (0.1591)

5. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE was considered related to the investigational drug product. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life -threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.TEAEs were defined as AEs/SAEs that started or worsened after the study drug treatment.
Time Frame: From the start of study drug administration up to Week 17
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Maralixibat 14 mcg/kg/Day: Participants received 14 mcg/kg/day of maralixibat oral solution for 1 week. One participant assigned to the 70μg/kg/day arm, was withdrawn from the study after receiving a single dose of 14 mcg/kg/day dose. TEAE was reported separately for this participant using this arm.
Arm/Group | Maralixibat 14 mcg/kg/Day | Maralixibat 70 mcg/kg/Day | Maralixibat 140 mcg/kg/Day | Maralixibat 280 mcg/kg/Day | Placebo
Number analyzed (Participants) | 1 | 7 | 11 | 6 | 12
Participants
  TEAE | 1 | 7 | 9 | 5 | 12
  Serious TEAE | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of study drug administration up to Week 17
Description: One participant assigned to the 70μg/kg/day arm, was withdrawn from the study after receiving a single dose of 14 mcg/kg/day dose. TEAE was reported separately for this participant in a separate arm.
Arm/Group | Maralixibat 14 mcg/kg/Day | Maralixibat 70 mcg/kg/Day | Maralixibat 140 mcg/kg/Day | Maralixibat 280 mcg/kg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/7 | 0/11 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/7 | 0/11 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 1/1 | 7/7 | 9/11 | 5/6 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maralixibat 14 mcg/kg/Day (N=1) | Maralixibat 70 mcg/kg/Day (N=7) | Maralixibat 140 mcg/kg/Day (N=11) | Maralixibat 280 mcg/kg/Day (N=6) | Placebo (N=12)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maralixibat 14 mcg/kg/Day (N=1) | Maralixibat 70 mcg/kg/Day (N=7) | Maralixibat 140 mcg/kg/Day (N=11) | Maralixibat 280 mcg/kg/Day (N=6) | Placebo (N=12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Growing pains (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 6 (8)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth crowding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 2 (3) | 2 (5) | 3 (5)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acoustic stimulation tests abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-Glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Enuresis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin e deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.